CLINICAL TRIAL: NCT05378750
Title: Fluid Overload Management and Vascular Stiffness in Chronic Kidney Disease Patients With Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00108113
Record Dates: First submitted 2022-04-01; First posted 2022-05-18 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
Keywords: Fluid Overload; Vascular Stiffness; Chronic Kidney Disease
MeSH Terms: conditions — Hypertension; Edema; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Bio-impedance spectroscopy.
  Treatment algorithm for diuretic therapy.
  Interventions: Other: Diuretic algorithm
- Control group (No Intervention): No intervention.

INTERVENTIONS:
Other: Diuretic algorithm — Implementing diuretic algorithm
  Arms: Intervention group

SUMMARY:
This study aims to reduce fluid overload in order to control blood pressure of hypertensive CKD patients using bio-impedance assessment of fluid status and using a diuretic therapy algorithm.

DETAILED DESCRIPTION:
Hypertension is highly prevalent in individuals with chronic kidney disease (CKD). Gradual loss of kidney function is associated with sodium retention. This ultimately leads to fluid overload which has been associated with high blood pressure and heart failure in patients with CKD. In such cases, diuretics are prescribed to reduce fluid overload and thereby control blood pressure. In clinical practice, diuretics are mostly prescribed based on clinical assessment of fluid status (e.g. hypertension, shortness of breath, edema). Less often biomarkers are used like brain natriuretic peptide and bio-impedance spectroscopy. Nevertheless, uncontrolled hypertension is highly prevalent in CKD patients, and leads to accelerated decline in kidney function as well as to cardiovascular disease. Bio-impedance spectroscopy is an accurate tool to assess fluid overload in CKD patients. Accurate assessment of fluid overload and appropriate prescription of diuretics are two pivotal factors to control blood pressure ultimately leading to preservation of kidney function in patients with CKD and decreased cardiovascular risk. Fluid overload in CKD is well documented, however, there are no randomized controlled trials demonstrating that strict fluid overload control in CKD patients improves blood pressure and outcome. Therefore, this study aims to reduce fluid overload in order to control blood pressure of hypertensive CKD patients using bio-impedance assessment of fluid status and using a diuretic therapy algorithm. First, fluid status will be assessed in all study participants using bio-impedance spectroscopy. Second, the study participants will be divided into two groups; the control group which will initially receive standard conventional therapy (no intervention) for 6 months. In the intervention group, the treatment regimen will be adjusted using bio-impedance spectroscopy and a treatment algorithm for diuretic therapy. Medications will be adjusted for 3 months and patients will be followed up for another 3 months. After 6 months, the control group will be subjected to the fluid overload management strategy. The primary outcomes of the current study are improvement in, a) fluid status towards normovolemia, and b) blood pressure toward normotension. Secondary outcome is improvement in vascular health as assessed by pulse wave velocity and augmentation index. Altogether, an optimized fluid status via a fluid management plan will provide better control of fluid overload, blood pressure, and improvement in vascular health in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old) outpatient with uncontrolled hypertension; defined as, AMBP ≥ 130/80 mmHg despite treatment
* With an estimated glomerular filtration rate (eGFR) of 15-45 ml/min/1.73 m2.
* Fluid overload of more than 5% of estimated normal ECFV, as assessed by Bio-impedance spectroscopy (we are using the Body Composition Monitor, a validated device marketed by Fresenius, Canada).

Exclusion Criteria:

* Pregnancy or lactation
* Declined informed consent
* Patients with cognitive dysfunction
* Surgery within six weeks of the study
* Patients with heart failure, atrial fibrillation, stroke, nephrotic syndrome and active auto-immune disease
* Patients with severe life-limiting comorbidities like cancer
* Patients with amputated limbs (despite the fact that the BCM device can be used if people have a unilateral amputation, the home devices measure via 2 legs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Fluid status | 12 months
  Decrease in fluid status measured using bio-impedance spectroscopy
Blood pressure | 12 months
  Decrease in blood pressure

SECONDARY OUTCOMES:
Vascular stiffness | 12 months
  Improvement in vascular health as assessed by augmentation index.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided